CLINICAL TRIAL: NCT02511665
Title: METformin And Longevity (METAL): A Window of Opportunity Study Investigating Biological Effects of Metformin in Localised Prostate Cancer
Brief Title: Metformin And Longevity
Acronym: METAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: METAL
Record Dates: First submitted 2015-07-27; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metformin (Experimental): Metformin given , 1g twice a day for 4 weeks until prostatectomy +/- one week
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): placebo given , 1g twice a day for 4 weeks until prostatectomy +/- one week
  Interventions: Drug: Placebo
- PET-MRI (Experimental): 5 patients in this arm will all receive metformin and undergo two additional PET- MRI scans, one before and one after treatment
  Interventions: Radiation: PET-MRI Scan

INTERVENTIONS:
Drug: Metformin — Given metformin
  Other Names: Glucophage
  Arms: Metformin
Radiation: PET-MRI Scan — Patients will under go 2 PET-MRI scans in the PET-MRI substudy arm one before treatment with metformin and one after
  Arms: PET-MRI
Drug: Placebo — Given placebo
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind, window of opportunity study investigating the biological mechanism of metformin in prostate cancer.

DETAILED DESCRIPTION:
A potential role for metformin in prostate cancer has been suggested and given its wide availability, tolerable side effect profile and safety record it may represent a therapeutic option for men with prostate cancer. However, the mechanism of action by which metformin exerts its anti-cancer effect has yet to be fully characterised. This 'window of opportunity' trial provides an opportunity to investigate this by comparing baseline prostate biopsies with post-treatment surgical specimen by focussing on assessment of the FASN/AMPK axis.

Patients with newly-diagnosed, early stage, prostate cancer scheduled for radical prostatectomy will either enter the main study and be randomised 1:1 to receive metformin (2g daily over 2 divided doses; Arm A) or placebo four weeks prior to prostatectomy (standard of care; Arm B). Or a subset of five patients will enter the exploratory PET-MRI Substudy . These five patients will all receive metformin and will undergo an additional two PET-MRI Scans.

Prostate tissue (at baseline from biopsy and post treatment from prostatectomy) will be used for analysis of p-AMPK, p-ACC, FASN by immunohistochemistry and proliferation will be measured using Ki67 and TUNEL in both metformin and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older and willing and able to provide signed informed consent.
2. Histologically confirmed adenocarcinoma of the prostate , with a minimum maximal tumour length of greater than 6mm on core biopsy
3. No previous treatment for prostate cancer (including surgery, any hormone therapy, radiotherapy and cryotherapy)
4. Prostate biopsy within 8 weeks from screening which contains sufficient material for baseline molecular marker assessment at Guy's and St Thomas' NHS Foundation trust..
5. Radical prostatectomy is the scheduled treatment of choice
6. Eastern Cooperative Oncology Group (ECOG) Performance status less than or equal to 0 or 1.
7. Adequate organ function, defined as follows:

   * Haemoglobin >10.0g/dL
   * Absolute neutrophil count >1.5x109/L
   * Platelet count >100x109/L
   * Renal function, eGFR >60ml/min (calculated by Cockcroft Gault)
   * AST and/or ALT <2.5 x ULN
   * Total Bilirubin <1.5 x ULN
8. Able to swallow the drug and comply with study requirements.

Exclusion Criteria:

1. Patients with a current or historical diagnosis of type one or two Diabetes and/or have ever received metformin
2. Patients with hypersensitivity to any of the components of Metformin or placebo tablet
3. History of or conditions associated with lactic acidosis such as shock or pulmonary insufficiency, alcoholism (acute or chronic), and conditions associated with hypoxaemia
4. Patients with chronic liver disease, severe cardiovascular impairment, cardiac failure, recent myocardial infarction, severe peripheral vascular disease or renal impairment (eGFR <60ml/min as measured by Cockcroft Gault)
5. Patients with acute severe disorders, for example infections with fever, pancreatitis, trauma, dehydration or reduced diet (<1000kcal or 4200kJ per day)
6. Other active malignancy over the last five years that has required systemic therapy, excluding:

   * Adjuvant therapy in the curative setting
   * Non-melanoma skin cancer
   * Superficial transitional cell carcinoma (CIS-T1)
7. Current enrolment in an investigational drug or device study or participation in such a study within 30 days of signing consent.
8. Any subjects who is able to father a child and does not agree to use barrier protection, in the form of a condom ,for the duration of the trial and for 16 weeks after the last study drug administration.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of the difference in expression levels of markers of the FASN/AMPK pathway pre and post treatment between the placebo and metformin arms. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rudman, MBBS BSc PhD, Principal Investigator — Guy's and St Thomas NHS Trust
Locations (1):
- Guy's Hospital, London, United Kingdom